CLINICAL TRIAL: NCT05448950
Title: Continued Access Study of the InterGraft™ Venous Anastomotic Connector for Minimally Invasive Connection of an Arteriovenous Graft for Hemodialysis
Brief Title: Continued Access Study VIG Anastomotic Connector
Acronym: VIG-CAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phraxis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIG-Continued Access Study
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Dialysis Access Malfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- VIG Continued Access (Experimental): Patients referred for AVG implant should be screened for study eligibility. A member of the Research Team will evaluate the patient for eligibility. If all initial inclusion criteria are met and no exclusion criteria are present, a member of the Research Team should inform the patient about the study's purpose and should obtain written informed consent.
  Final enrollment eligibility is determined at the time of surgery, after the physician has confirmed the final inclusion criterion is met. Enrolled subjects will be assigned a unique study subject identification number.
  Interventions: Device: VIG Continued Access Study

INTERVENTIONS:
Device: VIG Continued Access Study — Small skin incisions will be made for tunneling the graft under the skin in a standard manner. The VIG device is provided pre-loaded within a customized catheter-based delivery system for over-the-wire delivery. The VIG is inserted through an introducer sheath placed in the target vein so that the 'vessel end' of the VIG is deployed within the vein, and the 'graft end' extends out of the vein for connection to the graft. Delivery and deployment will be performed under fluoroscopic guidance. The VIG will be deployed first, connected to the AVG, then the graft and VIG will be flushed and clamped. The arterial anastomosis will then be created using a standard suturing method.
  Other Names: VIG Implant

SUMMARY:
The continued access study of the InterGraft Venous Anastomotic Connector (Venous InterGraft Continued Access Study, or 'VIG-CAS') allows for continued enrollment of subjects while the marketing application is being prepared and subsequently reviewed by FDA. The VIG-CAS will include the same patient population, follow-up schedule, and study endpoints as the VIG pivotal study.

DETAILED DESCRIPTION:
The VIG-CAS is a multicenter, prospective, single-arm study that will include up to 15 subjects contributed from up to 5 study sites that previously participated in the VIG pivotal study. No new investigators will be included. All subjects will be assigned to treatment with the VIG and a standard sutured arterial anastomosis for implantation of an arteriovenous graft (AVG) for hemodialysis. The selection criteria (patient population), follow-up schedule, and study endpoints are the same as those used in the pivotal study.

Study data will be collected up to the point at which each subject has completed the final 6-month follow up or experienced a terminal study event.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age.
2. Subject requires the creation of a vascular access graft for hemodialysis, secondary to a diagnosis of End Stage Renal Disease.
3. Subject has the vascular access graft placed in an upper extremity.
4. Baseline imaging shows suitable vascular anatomy/ vessel size for the InterGraft™ Venous Connector and an artery at least 3.5 mm in diameter that is suitable for creating the arterial anastomosis.
5. Subject has a reasonable expectation of remaining on hemodialysis for at least 6 months.
6. Subject or his/her legal guardian understands the study and is willing and able to comply with the dialysis schedule and follow-up requirements.
7. Subject or his/her legal guardian provides written informed consent. NOTE: In accordance with the requirements of some Institutional Review Boards (IRBs), where applicable, only those subjects with capacity to consent for themselves will be included. Thus, where required by the IRB, adult individuals who lack capacity to consent for themselves will be excluded from the study.
8. Physician's examination at time of surgery shows no significant vessel lesions, calcification(s), anatomic structures, or abnormalities that may limit ability to safely deploy the InterGraft™ Venous Connector or create a sutured arterial anastomosis.

Exclusion Criteria:

1. Subject has a documented and unsuccessfully treated ipsilateral central venous stenosis as determined by imaging.
2. Subject currently has a known or suspected bacterial, fungal, or HIV infection. NOTE: Subjects with hepatitis B or C may be included in the study.
3. Subject has a known hypercoagulable or bleeding disorder or requires treatment with warfarin or heparin. NOTE: The intent of this criterion is to exclude patients with high risk for bleeding or clotting complications. Patients who are taking the oral anticoagulant Eliquis® (apixaban) may be included in the study if Eliquis is temporarily discontinued prior to the study procedure, in accordance with the approved prescribing instructions. Patients may receive anticoagulation therapy any time after the study AV graft implant procedure, at their physician's discretion. This should be driven by an indication unrelated to the vascular access.
4. Subject has had a previous instance of Heparin Induced Thrombocytopenia type 2 (HIT-2) or has known sensitivity to heparin.
5. Subject has co-morbid conditions that may limit their ability to comply with study and follow-up requirements.
6. Subject has had >2 previous arteriovenous accesses in treatment arm.
7. Subject is currently taking Aggrenox®.
8. Subject needs or is scheduled for any major surgery within 30 days of the study procedure.
9. Subject is currently taking maintenance immunosuppressant medication such as rapamycin, mycophenolate or mycophenolic acid, prednisone (>10 mg), cyclosporine, tacrolimus, or cyclophosphamide.
10. Life expectancy is less than 12 months.
11. Subject is pregnant. NOTE: A negative urine pregnancy test within 24 hours of the study procedure is required in all female subjects with reproductive capacity.
12. Subject is a poor compliance risk (i.e.. history of IV or oral drug abuse).
13. Subject is enrolled in another dialysis or vascular investigational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Setum, PhD, Study Director — VP of Clinical Affairs
Locations (2):
- United States (2):
  - Trinity Research Group, LLC, Dothan, Alabama
  - Surgical Specialists of Charlotte, Charlotte, North Carolina

REFERENCES:
- [Background] Ebner A, Ross JR, Setum CM, Kallok MJ, Yevzlin AS. Transcatheter anastomosis connector system for vascular access graft placement: results from a first-in-human pilot study. J Vasc Access. 2016 Mar-Apr;17(2):111-7. doi: 10.5301/jva.5000481. Epub 2015 Oct 7. PMID 26450084
- [Background] Burgess JS, Beaver JD, London M, Rohan V, Orland P, Yevzlin A, Setum C, Ross J; InterGraft Study Investigators. Prospective multicenter study of a novel endovascular venous anastomotic procedure and device for implantation of an arteriovenous graft for hemodialysis. J Vasc Access. 2024 Jul;25(4):1244-1251. doi: 10.1177/11297298231159691. Epub 2023 Mar 9. PMID 36895157

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 patients were enrolled during June 7, 2022, to August 26, 2022. Although the study protocol allowed for enrollment of up to 15 patients, enrollment was stopped after 12 patients were enrolled, due to Sponsor decision to transfer the device to a new manufacturing facility.
Groups:
- VIG Continued Access: Patients referred for AVG implant were screened for study eligibility by a member of the research team. If all initial inclusion criteria were met and no exclusion criteria were present, the patient was informed of the study's purpose and invited to participate. Final enrollment eligibility was determined at the time of surgery, after the investigator confirmed the final inclusion criteria were met.
  Enrolled subjects were assigned a unique study subject identification number. Written informed consent was obtained from all enrolled patients prior to performing any study procedures.
  VIG Continued Access Study: Small skin incisions are made for tunneling the AVG under the skin in a standard manner. The VIG device is provided pre-loaded within a customized catheter-based delivery system for over-the-wire delivery. The VIG is inserted through an introducer sheath placed in the target vein so that the 'vessel end' of the VIG is deployed within the vein, and the 'graft end' extends out of the vein for manual insertion within the AVG. Delivery and deployment are performed under fluoroscopic guidance. The VIG is deployed first, connected to the AVG, then the AVG and VIG are flushed and clamped. The arterial anastomosis is then created using a standard suturing method.
Period: Overall Study
Arm/Group | VIG Continued Access
Started | 12
Completed | 5
Not Completed | 7
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1
Not completed — AVG abandoned | 4

BASELINE CHARACTERISTICS:
Arm/Group | VIG Continued Access
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 60.3 [35 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Diabetes mellitus [Count of Participants; unit: Participants] | 4
Obesity [Count of Participants; unit: Participants] | 2
Hypertension [Count of Participants; unit: Participants] | 12
Cardiovascular Disease [Count of Participants; unit: Participants] | 6
Hyperlipidemia [Count of Participants; unit: Participants] | 6
Current hemodialysis access using catheter [Count of Participants; unit: Participants] | 12
Location of implant VIG (and AVG) [Count of Participants; unit: Participants]
  left upper extremity | 5
  right upper extremity | 7

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Patency
Description: Percentage of subjects free from loss of access of the AVG for hemodialysis
Time Frame: 6 months
Population: Of 12 total enrolled subjects, 1 withdrew from the study before 6 months, after receiving a kidney transplant. Therefore, the number of subjects analyzed for the primary outcome measure is 11.
Measure: Count of Participants; unit: Participants
Arm/Group | VIG Continued Access
Number analyzed (Participants) | 11
Participants | 5

2. Secondary Outcome: Acute Device Success
Description: AVG flow at the end of the procedure as determined by palpable graft thrill and/or audible bruit, without significant bleeding or emergent surgery
Time Frame: At implant
Population: The analysis population includes all subjects that received the study device (all enrolled subjects).
Measure: Count of Participants; unit: Participants
Arm/Group | VIG Continued Access
Number analyzed (Participants) | 12
Participants | 12

3. Secondary Outcome: Primary Unassisted Patency
Description: Percentage of subjects free from the first occurrence of either access thrombosis or an access procedure performed to maintain access patency
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | VIG Continued Access
Number analyzed (Participants) | 11
Participants | 4

4. Secondary Outcome: Time to First Cannulation
Description: Time from initial access placement to the first graft cannulation for hemodialysis
Time Frame: 6 months
Measure: Mean (Full Range); unit: days
Arm/Group | VIG Continued Access
Number analyzed (Participants) | 12
days | 27.6 [9 to 50]

5. Secondary Outcome: Interventions Required to Maintain Secondary Patency
Description: Number and type of interventions required to maintain secondary patency. One or more intervention-types (e.g., angioplasty, thrombectomy, etc.) may have been performed during a single intervention surgery.
Time Frame: 6 months or up to time of early exit from the study, whichever occurs first.
Measure: Number; unit: Type of intervention
Units Other Than Participants: intervention surgeries
Arm/Group | VIG Continued Access
Number analyzed (Participants) | 12
Number analyzed (intervention surgeries) | 26
Type of intervention
  angioplasty | 12
  thrombectomy | 10
  thrombolytic infusion | 1
  stent placement | 3

6. Secondary Outcome: Protocol-defined Serious Adverse Events (SAEs)
Description: Protocol-defined SAEs (secondary endpoint) include the following: death, emergent surgery, AVG infection requiring treatment (e.g., prolonged or intravenous antibiotic therapy), significant bleeding (defined as bleeding requiring treatment), and pseudoaneurysm.
Time Frame: 6 months or up to time of early exit from the study, whichever occurs first.
Measure: Count of Participants; unit: Participants
Arm/Group | VIG Continued Access
Number analyzed (Participants) | 12
Participants
  Death | 2
  AVG infection | 1
  Emergent surgery | 0
  Significant bleeding | 0
  Pseudoaneurysm | 0
  No protocol-defined SAEs | 9

ADVERSE EVENTS:
Time Frame: Adverse event information was collected over a 6 month follow up period, or up to the date of a terminal study event (e.g., death, AVG abandonment, subject withdrawal), up to 6 months.
Arm/Group | VIG Continued Access
All-Cause Mortality (participants affected / at risk) | 2/12
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 4/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIG Continued Access (N=12)
pneumonia, requiring hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (2)
hematoma (Vascular disorders) | 1 (1) — Hematoma developed at needle puncture site (vascular access) on the AVG, causing damage to the AVG and necrosis in overlying skin. Treatment included excision of the mid-portion of the AVG.
cardiac arrest (Cardiac disorders) | 1 (1) — Subject had out of hospital cardiac arrest. CPR was provided and ROSC was obtained. Subject was transferred for comfort care, followed with subsequent death.
infection of AVG (Infections and infestations) | 1 (1)
abscess, tooth (Infections and infestations) | 1 (1) — abscess of tooth, subject hospitalized for treatment
cardiac arrest (Cardiac disorders) | 1 (1) — Subject had cardiac arrest while receiving hemodialysis. Despite resuscitation efforts, death occurred.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIG Continued Access (N=12)
pain (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) — The study protocol required that subjects with positive COVID-19 test be reported as an AE.
inflammation (General disorders) | 1 (1) — inflammation/redness at surgical incision site for AVG placement.
cancer, skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
bruising following a fall (General disorders) | 1 (1)
bleeding, minor (General disorders) | 1 (1) — minor bleeding at skin (incision) edge following AVG implantation procedure

LIMITATIONS AND CAVEATS:
Enrollment terminated early due to Sponsor's transfer of device manufacturing to a new facility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement states the following:

Research results and associated data generated by this Study conducted under this Agreement will be considered confidential until the first publication or presentation thereof of data according to the terms of this Agreement or one (1) year after conclusion, abandonment or termination of the Study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT05448950/Prot_SAP_000.pdf